CLINICAL TRIAL: NCT02611661
Title: Local Ablative Strategies After Endovascular Radioembolization (LASER)
Brief Title: Local Ablative Strategies After Endovascular Radioembolization
Acronym: LASER
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Principal Investigator left the university.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201511087
Record Dates: First submitted 2015-11-18; First posted 2015-11-23 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Catheter Ablation; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- Stratum 1: Observe (Other): * PET/MRI within 36 hours of standard of care hepatic radioembolization received off study
  * No further treatment just observation
  Interventions: Device: PET/MRI
- Stratum 2: Percutaneous ablation (Experimental): * PET/MRI within 36 hours of standard of care hepatic radioembolization received off study
  * Percutaneous ablation can be radiofrequency ablation (RFA), microwave ablation (MWA), cryoablation, and irreversible electroporation
  Interventions: Device: PET/MRI; Radiation: Percutaneous ablation
- Stratum 3: SBRT (Experimental): * PET/MRI within 36 hours of standard of care hepatic radioembolization received off study
  * The planned SBRT dose will be 30 Gy in 5 fractions of 6 Gy each. It is recommended that each fraction be separated by a minimum of 12 hours and a maximum of 8 days.
  Interventions: Device: PET/MRI; Radiation: Stereotactic body radiotherapy
- Stratum 4: SBRT + Percutaneous Ablation (Experimental): * PET/MRI within 36 hours of standard of care hepatic radioembolization received off study
  * Percutaneous ablation can be radiofrequency ablation (RFA), microwave ablation (MWA), cryoablation, and irreversible electroporation
  * The planned SBRT dose will be 30 Gy in 5 fractions of 6 Gy each. It is recommended that each fraction be separated by a minimum of 12 hours and a maximum of 8 days.
  Interventions: Device: PET/MRI; Radiation: Percutaneous ablation; Radiation: Stereotactic body radiotherapy
- Stratum 5: Referral for systemic therapy (No Intervention): * PET/MRI within 36 hours of standard of care hepatic radioembolization received off study
  * Referred for further systemic therapy and are not candidates for further locoregional therapy on study.

INTERVENTIONS:
Device: PET/MRI
  Arms: Stratum 1: Observe; Stratum 2: Percutaneous ablation; Stratum 3: SBRT; Stratum 4: SBRT + Percutaneous Ablation
Radiation: Percutaneous ablation
  Arms: Stratum 2: Percutaneous ablation; Stratum 4: SBRT + Percutaneous Ablation
Radiation: Stereotactic body radiotherapy
  Other Names: SBRT
  Arms: Stratum 3: SBRT; Stratum 4: SBRT + Percutaneous Ablation

SUMMARY:
The rationale for this design is initial utilization of a standard-of-care therapy for mCRC (radioembolization) with a dose-calculation algorithm that has been verified as predictive for treatment response. Prediction of treatment failure will enable the proposed subsequent locoregional therapies which were selected based on safety profiles and feasibility. While the goal of this study is assessing feasibility and safety of this approach, the end goal of improving overall patient outcomes by improved hepatic tumor control.

DETAILED DESCRIPTION:
As the median time to radiographic response ranges from 3-8 months in published data, utilization of post-treatment PET/MRI dosimetry offers a powerful mechanism for immediate (within 36 hours) prediction of lesions that are likely to fail radioembolization. This early prediction enables a window for subsequent locoregional therapy prior to re-initiation of systemic chemotherapy. The investigators propose to evaluate patients who are undergoing radioembolization for mCRC using PET/MRI derived dosimetry obtained within 36 hours of the radioembolization procedure. Patients with four tumors or fewer receiving an average dose (Davg) less than 30 Gy will be candidates for subsequent locoregional therapy (stereotactic body radiotherapy (SBRT) or microwave ablation). This strategy will ideally increase the therapeutic index of locoregional therapies, particularly in the patient population who has exhausted their options for systemic therapy.

After radioembolization, patients will be divided into 5 strata as per the protocol schema. Patients who receive a Davg greater than 30 Gy in all hepatic lesions will be placed in Stratum 1 and will not undergo subsequent therapy. Patients with four or fewer lesions receiving a Davg less than 30 Gy will be placed in Strata 2, 3, or 4 based on distribution of the underdosed lesions. Stratum 2 will be comprised of patients with four or fewer underdosed lesions less than 3 cm which do not touch vasculature greater than 4 mm in size. Patients in this stratum will receive percutaneous microwave ablation to the underdosed lesions. Stratum 3 will be composed of patients with 4 or fewer underdosed lesions that are not amenable to microwave ablation by virtue of either size (greater than 3 cm) or proximity to hepatic vasculature greater than 4 mm in diameter. These patients will be treated with SBRT to the underdosed lesions. Patients with a combination of lesions some of which are amenable to microwave ablation and some of which are not (due to either size or proximity to vasculature) will be treated in Stratum 4 with a combined approach - microwave ablation to all lesions which are amenable and SBRT to any remaining underdosed lesions. Finally, Stratum 5 will consist of patients with more than 4 underdosed lesions or with disease progression; these patients will be referred for further systemic therapy and are not candidates for further locoregional therapy on study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of colorectal carcinoma with intrahepatic metastases; limited extrahepatic metastasis is allowed as long as the overall metastatic burden is hepatic dominant.
* Local surgical resection is not possible due to tumor or patient factors.
* Prior locoregional therapy is allowed if completed at least 2 weeks prior to enrollment.
* Prior chemotherapy is allowed if stopped/completed at least 2 weeks prior to enrollment.
* At least 18 years old.
* ECOG performance status ≤ 1.
* Scheduled to undergo radioembolization for treatment of intrahepatic metastases.
* Able to understand and willing to sign an IRB-approved written informed consent document.

Exclusion Criteria:

* Child-Pugh score 8 or greater.
* ALT or AST ≥ 6 x ULN.
* Prior history of abdominal irradiation. Patients who have received prior pelvic radiation for colorectal cancer are eligible; however, prior radiation treatment plans must be reviewed prior to enrollment.
* Presence of any contraindications to MRI scanning.
* GFR < 30 ml/min/1.73m2 (if receiving contrast for MRI).
* Currently on dialysis (if receiving contrast for MRI).
* Prior allergic reaction to gadolinium-based contrast agents (if receiving contrast for MRI).
* Pregnant or nursing. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-01-19 (Actual); Primary Completion 2018-02-13 (Actual); Study Completion 2018-02-13 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of administering hepatic locoregional therapy following radioembolization as measured by occurrences of grade 3 or higher toxicities of interest | 30 days after completion of therapy (approximately 6 weeks)
  * Strata 2, 3, and 4 only
  * The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.

SECONDARY OUTCOMES:
Late toxicity associated with radioembolization followed by dosimetry-guided subsequent hepatic locoregional therapy | Up to 6 months
  -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.
Local recurrence rates associated with radioembolization followed by dosimetry-guided subsequent hepatic locoregional therapy | Up to 2 years
Overall survival rates associated with radioembolization followed by dosimetry-guided subsequent hepatic locoregional therapy | Up to 2 years
Response rates associated with radioembolization followed by dosimetry-guided subsequent hepatic locoregional therapy | Up to 6 months
  * Complete Response (CR): Disappearance of all target lesions and non-target lesions. Normalization of tumor marker level.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  * Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
  * Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.

CONTACTS AND LOCATIONS:
Overall Officials: Parag Parikh, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu